CLINICAL TRIAL: NCT06183359
Title: Correct Self-identification Program in the Treatment of Depression: a Randomized Controlled Trial
Brief Title: Self-Identification Program
Acronym: SIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL21_0280
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder; Third Wave Cognitive Behavioral Therapy
Keywords: Depression; psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: The group Self-Identification Program (SIP) versus The group Acceptance and Commitment Therapy (ACT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group Self-Identification Program (SIP) (Experimental): The Self-Identification Program (SIP) is a third level of third wave CBT.
  It targets a correct self-identification through the of the following skills :
  * understand the nature and functioning of one's own mind (=conscious power, what allows the appearance of experiences);
  * learn to identify with the characteristics of the mind : to provide soothing (session 1), reassuring power (session 2), benevolent power (session 3), discerning power (session 4), prioritizing power (session 5), acting power (session 6), creative power (session 7), liberating power (session 8)
  * live better with your emotions and moods (and their dysregulation);
  * develop more respectful communication for oneself and others
  Interventions: Other: SIP
- The group Acceptance and Commitment Therapy (ACT) (Other): The Acceptance and Commitment Therapy (ACT) is a first level of third wave CBT.
  It targets the development of the following skills, consistent with the content of programs validated in the domain :
  * decision-making tool (matrix (session 1));
  * flexibility skills: defusion (session 2), Self as context (session 4), acceptance (session 4), contact with the present moment (session 5), values (session 6), valued actions (session 7), toolkit skills (session 8).
  Interventions: Other: SIP

INTERVENTIONS:
Other: SIP — compare the SIP group versus the ACT group

SUMMARY:
Conduct a pilot, single-center, randomized controlled 2-arm study aimed to evaluate the impact of an in-depth 3rd wave CBT program targeting correct self-identification (3rd level of 3rd wave CBT), compared to a control group receiving an acceptance and commitment therapy (ACT; (1st level of 3rd wave CBT, a well-known psychotherapy). Main judgment criteria : Therapeutic response (reduction ≥ 50% between pre and immediate post-treatment), and rate of relapse at 6 months post-therapy. Secondary objectives: Evaluate psychological processes involved in the reduction of moral pain, diligence, ruminations, suicidal ideas, self-concept and alterations in functioning (mental and social), psychological skills.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), depression is one of the health problems most prevalent mental health issues of the 21st century. Currently available treatments are insufficient to treat effectively combat depression, prevent relapse, and provide a care offer accessible to all people. requiring. Self-identification is at the heart of the dimensional understanding of this disorder, including moral pain inherent is associated with excess suicide mortality. From altered relationships to negative affectivity and affectivity positive are central psychological processes that maintain depression and promote relapse. Cognitive and behavioral psychotherapies (CBT) are the reference in addition to medications. The paramedical team (nurses and psychologists) of the Therapies Center (CHU Montpellier) has created a program targeting correct Self-Identification (SIP; 3rd level of 3rd wave CBT), allowing the reestablishment of functional relationships. This notable innovation was welcomed by the World Health Organisation, which requested its presentation during the meeting of the United Nations in Geneva in June 2021 (international exhibition on resilience).

Main objectives: Conduct a pilot, single-center, randomized controlled 2-arm study aimed to evaluate the impact of an in-depth 3rd wave CBT program targeting correct self-identification (3rd level of 3rd wave CBT), compared to a control group receiving an acceptance and commitment therapy (ACT; (1st level of 3rd wave CBT, a well-known psychotherapy). Main judgment criteria : Therapeutic response (reduction ≥ 50% between pre and immediate post-treatment), and rate of relapse at 6 months post-therapy. Secondary objectives: Evaluate psychological processes involved in the reduction of moral pain, diligence, ruminations, suicidal ideas, self-concept and alterations in functioning (mental and social), psychological skills.

Statistical analysis: A descriptive analysis of the initial characteristics of the patients will be carried out in each of the groups to check initial comparability. The analyzes of the judgment criteria will be carried out with an intention-to-treat analysis.

Feasibility: Paramedical team (nurses and psychologists) specialized in 3rd wave CBT (200 patients/week), coordinated by Dr Ducasse (internationally recognized in the field).

Outcomes/prospects: This program should 1) reduce the frequency and intensity of mental illnesses symptoms, and the associated mental pain, 2) prevent the negative consequences of mental illnesses (poor quality of life, isolation, self-damaging behavior), 3) reduce the mental illness stigma.

3rd wave CBTs constitute programs that can be delivered in group sessions by both nurses and psychologists, with appropriate training. This ensures its potential for wide distribution, where France faces a shortage of psychotherapeutic offerings.

Such a program will undeniably constitute an important contribution on the dimensional understanding of mental illnesses, and the implementation of innovative transnosographic psychotherapeutic care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years, presenting a current major depressive episode (according to DSM 571), as part of unipolar or bipolar depressive disorder

Exclusion Criteria:

* Patients with a psychotic disorder
* Patients with active thoughts of suicide with intention to carry out the act (C-SSRS "ideation suicidal" in the last week ≥ 4)
* Inability to receive informed information about the study
* Exclusion period determined by a previous study
* Adult protected by law or patient under guardianship or curatorship
* Not be affiliated to a French social security scheme or beneficiary of such a scheme
* Not being able to give informed written consent
* Pregnant or breastfeeding women
* Patients under judicial protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) | Between pre- and immediate post-therapy, 3 months post-intervention and 6 months after the intervention (in the intervention group compared to the control group)
  Depressive symptomatology

SECONDARY OUTCOMES:
montgomery asberg depression scale (MADRS) | Between pre- and immediate post-therapy, 3 months post-intervention and 6 months after the intervention (in the intervention group compared to the control group)
  Depressive symptomatology
Variation in moral pain | Between pre- and immediate post-therapy, 3 months post-intervention and 6 months after the intervention (in the intervention group compared to the control group)
  visual analog scale 0-10
Functioning Assessment Short Test (FAST) | Between pre- and immediate post-therapy, 3 months post-intervention and 6 months after the intervention (in the intervention group compared to the control group)
  Overall functionning
Columbia-Suicide Severity Rating Scale (C-SSRS) | Between pre- and immediate post-therapy, 3 months post-intervention and 6 months after the intervention (in the intervention group compared to the control group)
  Suicidal behaviors
anxious symptomatology (STAI-State) | Between pre- and immediate post-therapy, 3 months post-intervention and 6 months after the intervention (in the intervention group compared to the control group)
  anxious symptomatology
Snaith-Hamilton Pleasure Scale (SHAPS) | Between pre- and immediate post-therapy, 3 months post-intervention and 6 months after the intervention (in the intervention group compared to the control group)
  Anhedonia

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No